CLINICAL TRIAL: NCT03703362
Title: Resistance Training for Patients Diagnosed With External Snapping Hip. A Feasibility Study
Brief Title: Resistance Training for Patients Diagnosed With External Snapping Hip
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SnappingHip
Record Dates: First submitted 2018-05-29; First posted 2018-10-11 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2018-05

CONDITIONS: Coxa Saltans External
Keywords: Resistance training; Feasibility
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Progressive resistance training (Experimental): Progressive resistance training tested in patients with external snapping hip
  Interventions: Other: Resistance training

INTERVENTIONS:
Other: Resistance training — 30 supervised training-sessions over 12 weeks

SUMMARY:
The purpose of this study is to investigate whether targeted progressive resistance training is safe and feasible for patients with external snapping hip. Dropout rates, adverse events and training adherence are investigated. The secondary purpose is to investigate whether it is possible through targeted progressive resistance training to improve participants' muscle strength, functional status and hip-related quality of life.

DETAILED DESCRIPTION:
Snapping hip (coxa saltans) is a disorder where the hip tends to make an audible click-through movement, often but not necessarily associated with pain. A prevalence of 5-10% of the general population has been reported. Snapping hip is divided into three forms of snapping hip; intraarticular, internal and external snapping hip. External snapping hip (coxa saltans external) is the most common form, and patients may experience pain when the iliotibial band or anterior part of the gluteus maximus slides over the greater trochanter at femur. Patients with external snapping hip are typically between 15 and 40 years, and physically active.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Greater Trochanteric Pain Syndrome at the Orthopedic Surgery Department at Aarhus University Hospital in the period 2013-2015. In case of too few participants from this sample, we plan to include patients diagnosed during 2018
* Minimum 18 years old
* Able to read and understand Danish
* Have experienced jump/click from the outside of the hip associated with pain within the last 14 days
* Have a residence of a maximum of 55 km from Aarhus C
* The participants must not have participated in regular resistance training of the hip muscles for more than 1 day per week in the last 6 months leading up to the start of the intervention
* The participants must not have undergone a total hip replacement, a Periacetabular Osteotomy, a Z-plastic surgery or arthroscopy in the hip within 6 months before the start of the intervention or have a planned hip surgery during the intervention period
* The participants must not suffer from neurological, rheumatological, metabolic or respiratory diseases that will influence the effect of the intervention
* The participants must not have a planned vacation lasting more than 14 days during the intervention period, while not having the opportunity to extend the training period accordingly

Exclusion Criteria:

* BMI >40
* No longer suffering from external snapping hip
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2019-03-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Adverse events. | Measured at each training session during the 12 week intervention.
  A muscle or joint injury caused by the training program reported by a patient, or a canceled training session due to pain associated with exercise, or other harmful incidents associated with the training program.
Pain during exercise. | Measured for each exercise performed during the 12 week intervention.
  Pain during the exercises, measured by the Visual Analogue Scale (VAS). The score range from 0-10, where 0 means no pain and 10 means maximum pain
Adherence to the training. | Measured during the 12 week intervention.
  Measured by how many of the training sessions the participants completed. High adherence defined >80% of completed sessions. Drop out is defined as a person included in the study who chooses to leave before the final test.

SECONDARY OUTCOMES:
Change in muscle strength measured by dynamometer. | Measured at inclusion, two weeks after inclusion, and when the 12 week intervention has ended.
  Muscle strength in hip-abduction and hip-extension is measured isometrically, eccentrically and concentrically with a dynamometer (model Humac Norm).
Change in hip function. | Measured at inclusion, two weeks after inclusion, and when the 12 week intervention has ended.
  Hip function is measured with the questionnaire the Copenhagen Hip and Groin Outcome Score (HAGOS). HAGOS consists of 37 items in 6 subscales: 7 items to cover symptoms, 10 items to cover pain, 5 items to cover physical function in daily living, 8 items to cover physical function in sport and recreation, 2 items to cover participation in physical activities and 5 items to cover hip and groin related quality of life. There is no total score. Each subscale has a range from 0-100. A high score indicates no problem and a low score indicates severe problems.
Hypermobility status. | Measured at inclusion, two weeks after inclusion and when the 12 week intervention has ended.
  Hypermobility status is measured with the Beighton Score. The test consists of 9 activities and each of the 9 tests can result in a score of 0 or 1 depending on whether the patient can perform the test or not. A total score is summed and has a range of 0-9. Hypermobility is defined by a score of 5 or higher.
Change in one repetition muscle strength. | At the start of the intervention and 12 weeks later at the end of the intervention.
  Muscle strength is measured with the One-Repetition-Max test for hip-abduction and leg press.
Change in hip function. | Measured at inclusion, two weeks after inclusion and when the 12 week intervention has ended.
  Change in hip function is measured with a Loaded stair test.
Hip awareness. | Measured at inclusion, two weeks after inclusion and when the 12 week intervention has ended.
  Hip awareness is measured with the Forgotten Joint Score questionnaire (FJS), where each patient completes the 12 questions regarding awareness of their affected hip. Each question is answered with one of the following options; never, almost never, seldom, sometimes and mostly, corresponding to a score of 1-5. The sum of the scores will be converted into a score between 0-100. A high score will indicate lack of awareness and a low score will indicate great awareness of the affected hip.

CONTACTS AND LOCATIONS:
Overall Officials: Inger Mechlenburg, Study Director — Aarhus University Hospital
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Aarhus
  - Horsens Regional Hospital, Horsens
  - Silkeborg Regional Hospital, Silkeborg